CLINICAL TRIAL: NCT03323567
Title: A Comparison of Collagen, Lidocaine and Saline Intramuscular Injections, in Myofascial Pain Patients With Trigger Points in Masseter Muscle.
Brief Title: A Comparison of Collagen, Lidocaine and Saline, in Trigger Points in Masseter Muscle.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Aleksandra Nitecka-Buchta, Principal Investigator D.M.D. PhD, Medical University of Silesia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Silesian UM
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Temporomandibular Disorder
Keywords: TMD, collagen, intramuscular injection, trigger point
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Lidocaine; Injections; Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: patients were divided into the three groups and examination and therapy was performed after 7 and 14 days
Who Masked: Participant, Care Provider
Masking Description: Participants and care providers had no knowledge about the substance prepared for the injection. The information for the main investigator was the number of patient and the number of injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (3):
- MD Muscle Collagen group (Experimental): Group with collagen intramuscular injections
  Interventions: Drug: MD Muscle GUNA collagen
- Lidocaine 2% group (Experimental): Group with 2% Lidocaine intramuscular injections
  Interventions: Drug: Lidocaine 2% Injectable Solution
- Saline (Placebo Comparator): Group with 0,9% NaCl intramuscular injections
  Interventions: Drug: Saline Solution, Hypertonic

INTERVENTIONS:
Drug: MD Muscle GUNA collagen — intramusclular injections of MD Muscle collagen
  Other Names: intramuscular MD Muscle collagen injection
  Arms: MD Muscle Collagen group
Drug: Lidocaine 2% Injectable Solution — intramuscular Lidocaine 2% injection
  Other Names: intramuscular Lidocaine 2% injection
  Arms: Lidocaine 2% group
Drug: Saline Solution, Hypertonic — intramuscular Saline injection
  Other Names: intramuscular Saline injection
  Arms: Saline

SUMMARY:
An intramusclular injection of three solutions were performed( collagen, lidocaine, saline) in musculoskeletal trigger points, in patients suffering from temporomandibular disorders(TMD). Best results were observed in collagen group: reduction of 59,2% sEMG activity of masseter muscles and 53,75% reduction of pain intensity in VAS scale.

DETAILED DESCRIPTION:
Collagen is an important component, building myocytes and extracellular matrix of skeletal muscles. The novel treatment option for trigger point therapy and muscle regeneration in TMD patients are intramuscular collagen injections. The aim of the study was to evaluate the efficacy of intramuscular injections of Collagen MD Muscle(Guna) 2 ml, 2 ml of Lidocainum 2% without vasoconstrictor and 2 ml of Saline (0,9 % NaCl). 43 patients were enrolled to the study (17 male and 26 female, 40 +/- 3,8 years old). The masseter muscle activity was measured with sEMG Neurobit Optima 4 (Neurobit System). Visual Analogue Scale was used to determine pain intensity changes between follow-up visits in each group. Trigger points were localized with palpation of masseter muscle. Electromyographic activity of masseter muscle was measured before injections on each visit: 0, 7,14 days. In our analysis sEMG masseter muscle activity was significantly decreased: in collagen group 59,2%, in lidocainum group 39,3% and in saline group14%. Pain intensity reduction in VAS scale was 53,75% in collagen group, in lidocainum group 25% and in saline group 20,1%.

ELIGIBILITY:
Inclusion Criteria:

- sleep bruxism, DC/TMD myofascial pain, myofascial pain with referral

Exclusion Criteria:

* younger than 18years old, active orthodonctic treatment,neurological treatment, post radiotherapy, after head trauma within 2 years, patients with unsupported occlusal contacts, addicted to analgesic drugs, with the fear of needle

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-01-10; Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
sEMG reduction of masseter muscle in TMD patients | 14 days
  reduction of electromyograpic activity of masseter muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Department of TMD and Orthodontics Silesian Medical University, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Turo D, Otto P, Hossain M, Gebreab T, Armstrong K, Rosenberger WF, Shao H, Shah JP, Gerber LH, Sikdar S. Novel Use of Ultrasound Elastography to Quantify Muscle Tissue Changes After Dry Needling of Myofascial Trigger Points in Patients With Chronic Myofascial Pain. J Ultrasound Med. 2015 Dec;34(12):2149-61. doi: 10.7863/ultra.14.08033. Epub 2015 Oct 21. PMID 26491094
- [Background] Jarvholm U, Palmerud G, Styf J, Herberts P, Kadefors R. Intramuscular pressure in the supraspinatus muscle. J Orthop Res. 1988;6(2):230-8. doi: 10.1002/jor.1100060210. PMID 3343629
- [Background] Lehto M, Sims TJ, Bailey AJ. Skeletal muscle injury--molecular changes in the collagen during healing. Res Exp Med (Berl). 1985;185(2):95-106. doi: 10.1007/BF01854894. PMID 3992061
- [Background] Sorichter S, Mair J, Koller A, Gebert W, Rama D, Calzolari C, Artner-Dworzak E, Puschendorf B. Skeletal troponin I as a marker of exercise-induced muscle damage. J Appl Physiol (1985). 1997 Oct;83(4):1076-82. doi: 10.1152/jappl.1997.83.4.1076. PMID 9338413
- [Background] Cescon M, Gattazzo F, Chen P, Bonaldo P. Collagen VI at a glance. J Cell Sci. 2015 Oct 1;128(19):3525-31. doi: 10.1242/jcs.169748. Epub 2015 Sep 16. PMID 26377767
- [Derived] Nitecka-Buchta A, Walczynska-Dragon K, Kempa WM, Baron S. Platelet-Rich Plasma Intramuscular Injections - Antinociceptive Therapy in Myofascial Pain Within Masseter Muscles in Temporomandibular Disorders Patients: A Pilot Study. Front Neurol. 2019 Mar 19;10:250. doi: 10.3389/fneur.2019.00250. eCollection 2019. PMID 30941095